CLINICAL TRIAL: NCT04727216
Title: Intermittent Dorsal Root Ganglion Stimulation Dosing Comparison to Standard Continuous Dosing in Treating Chronic Pain
Brief Title: Intermittent vs. Continuous Dorsal Root Ganglion Stimulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spine and Pain Institute of New York (Other)
Responsible Party: Principal Investigator, Kenneth Chapman, Principle Investigator, Spine and Pain Institute of New York
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Intermittent DRG-S Dosing
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Pain, Intractable; Pain, Chronic
Keywords: Dorsal Root Ganglion Stimulation; Intermittent Stimulation Dosing
MeSH Terms: conditions — Pain, Intractable; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Subjects will undergo 3 sequential 2-week dosing stimulation programs [1.) continuous, 2.) 1 minute on: 1 minute off, and 3.) 1 minute on: 2 minutes] in randomized order and double blinded fashion for a total of 6 consecutive weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to which stimulation program they are receiving during each 2 week cycle. The Investigator who is also the care provider will be blinded to both the stimulation they are receiving and the sequential order they are given in. The outcomes assessor will be blinded to the sequential order of the stimulation programs each participant receives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Continuous DRG-S Dosing (Active Comparator): 2 week stimulation program using continuous DRG-S dosing at standard stimulation parameters
  Interventions: Device: Dorsal Root Ganglion Stimulation (DRG-S)
- 1 minute on: 1 minute off Intermittent DRG-S Dosing (Experimental): 2 week stimulation program using 1 minute on: 1 minute off intermittent DRG-S dosing at standard stimulation parameters
  Interventions: Device: Dorsal Root Ganglion Stimulation (DRG-S)
- 1 minute on: 2 minutes off Intermittent DRG-S Dosing (Experimental): 2 week stimulation program using 1 minute on: 2 minutes off intermittent DRG-S dosing at standard stimulation parameters
  Interventions: Device: Dorsal Root Ganglion Stimulation (DRG-S)

INTERVENTIONS:
Device: Dorsal Root Ganglion Stimulation (DRG-S) — Dorsal Root Ganglion stimulation will be delivered with continuous dosing and 2 different ON/OFF periods to compare effects for each patient.

SUMMARY:
The purpose of this study is to evaluate and compare the therapeutic efficacy of intermittent Dorsal Root Ganglion Stimulation (DRG-S) to standard continuous stimulation in patients with chronic intractable pain

DETAILED DESCRIPTION:
Intermittent Dorsal Root Ganglion Stimulation (DRG-S) dosing consists of preprogrammed cycles during which stimulation is delivered with standard DRG-S parameters alternated with periods during which no stimulation is being delivered.

In this study the investigators propose to evaluate therapeutic efficacy of Intermittent DRG-S at 1 minute on: 1 minute off and 1 minute on: 2 minute off dosing in comparison to standard continuous DRG-S dosing and determine if there is noninferiority between the intermittent and continuous paradigms in chronic pain patients with permanent DRG-S implants.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide informed consent to participate in the study;
* Subject is 21 years of age or older;
* Subject has been treated with DRG-S permanent implant device (Abbott, Plano, TX, USA) for a minimum of 3 months with sustained pain relief >50% for chronic intractable pain;
* Subject's DRG-S parameters have remained unchanged for at least 30 days prior to the beginning of the study

Exclusion Criteria:

* Subject had a recent change in pain medication regimen resulting in increase in Morphine Milligram Equivalent dosing within 60 days prior to the beginning of the study
* Subject received an additional pain interventional procedure within 60 days prior to the beginning of the study

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Numerical Rating Scale (NRS) Pain Scores Between Continuous and 1:1 Intermittent Dosing | After 2 weeks of continuous stimulation dosing and after 2 weeks of 1:1 intermittent dosing
  Pain Questionnaire - (Scale is 0 to 10 with 0 being no pain and 10 being worst pain imaginable)
Change in Numerical Rating Scale (NRS) Pain Scores Between Continuous and 1:2 Intermittent Dosing | After 2 weeks of continuous stimulation dosing and after 2 weeks of 1:2 intermittent dosing
  Pain Questionnaire - (Scale is 0 to 10 with 0 being no pain and 10 being worst pain imaginable)

SECONDARY OUTCOMES:
Change in Quality of Life Between Continuous and 1:1 Intermittent Dosing | After 2 weeks of continuous stimulation dosing and after 2 weeks of 1:1 intermittent dosing
  Questionnaire on quality of life using european quality of life - 5 dimension questionnaire (EQ-5D) - (Scale is between 0 and 1 with 0 being worse quality of life and 1 best quality of life)
Change in Quality of Life Between Continuous and 1:2 Intermittent Dosing | After 2 weeks of continuous stimulation dosing and after 2 weeks of 1:2 intermittent dosing
  Questionnaire on quality of life using european quality of life - 5 dimension questionnaire (EQ-5D) - (Scale is between 0 and 1 with 0 being worse quality of life and 1 best quality of life)
Change in Disability Index Between Continuous and 1:1 Intermittent Dosing | After 2 weeks of continuous stimulation dosing and after 2 weeks of 1:1 intermittent dosing
  Questionnaire on disability, Oswestry Disability Index (ODI) - (Scale is between 0 and 100 with 0 being no disability and 100 worst disability)
Change in Disability Index Between Continuous and 1:2 Intermittent Dosing | After 2 weeks of continuous stimulation dosing and after 2 weeks of 1:2 intermittent dosing
  Questionnaire on disability, Oswestry Disability Index (ODI) - (Scale is between 0 and 100 with 0 being no disability and 100 worst disability)

OTHER OUTCOMES:
Stimulation Program Peference | 6 week follow up visit after completing all 3 stimulation programs
  Percentage of patients preferring each stimulation program

CONTACTS AND LOCATIONS:
Locations (1):
- Spine and Pain Institute NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deer TR, Levy RM, Kramer J, Poree L, Amirdelfan K, Grigsby E, Staats P, Burton AW, Burgher AH, Obray J, Scowcroft J, Golovac S, Kapural L, Paicius R, Kim C, Pope J, Yearwood T, Samuel S, McRoberts WP, Cassim H, Netherton M, Miller N, Schaufele M, Tavel E, Davis T, Davis K, Johnson L, Mekhail N. Dorsal root ganglion stimulation yielded higher treatment success rate for complex regional pain syndrome and causalgia at 3 and 12 months: a randomized comparative trial. Pain. 2017 Apr;158(4):669-681. doi: 10.1097/j.pain.0000000000000814. PMID 28030470
- [Background] Miller JP, Eldabe S, Buchser E, Johanek LM, Guan Y, Linderoth B. Parameters of Spinal Cord Stimulation and Their Role in Electrical Charge Delivery: A Review. Neuromodulation. 2016 Jun;19(4):373-84. doi: 10.1111/ner.12438. Epub 2016 May 6. PMID 27150431
- [Background] Chapman KB, Yousef TA, Foster A, D Stanton-Hicks M, van Helmond N. Mechanisms for the Clinical Utility of Low-Frequency Stimulation in Neuromodulation of the Dorsal Root Ganglion. Neuromodulation. 2021 Jun;24(4):738-745. doi: 10.1111/ner.13323. Epub 2020 Nov 25. PMID 33236811
- [Background] Chapman KB, Yousef TA, Vissers KC, van Helmond N, D Stanton-Hicks M. Very Low Frequencies Maintain Pain Relief From Dorsal Root Ganglion Stimulation: An Evaluation of Dorsal Root Ganglion Neurostimulation Frequency Tapering. Neuromodulation. 2021 Jun;24(4):746-752. doi: 10.1111/ner.13322. Epub 2020 Nov 23. PMID 33227827
- [Background] Esposito MF, Malayil R, Hanes M, Deer T. Unique Characteristics of the Dorsal Root Ganglion as a Target for Neuromodulation. Pain Med. 2019 Jun 1;20(Suppl 1):S23-S30. doi: 10.1093/pm/pnz012. PMID 31152179
- [Background] Koopmeiners AS, Mueller S, Kramer J, Hogan QH. Effect of electrical field stimulation on dorsal root ganglion neuronal function. Neuromodulation. 2013 Jul-Aug;16(4):304-11; discussion 310-1. doi: 10.1111/ner.12028. Epub 2013 Feb 19. PMID 23421796
- [Background] Arcourt A, Gorham L, Dhandapani R, Prato V, Taberner FJ, Wende H, Gangadharan V, Birchmeier C, Heppenstall PA, Lechner SG. Touch Receptor-Derived Sensory Information Alleviates Acute Pain Signaling and Fine-Tunes Nociceptive Reflex Coordination. Neuron. 2017 Jan 4;93(1):179-193. doi: 10.1016/j.neuron.2016.11.027. Epub 2016 Dec 15. PMID 27989460
- [Background] Koetsier E, Franken G, Debets J, van Kuijk SMJ, Linderoth B, Joosten EA, Maino P. Dorsal Root Ganglion Stimulation in Experimental Painful Diabetic Polyneuropathy: Delayed Wash-Out of Pain Relief After Low-Frequency (1Hz) Stimulation. Neuromodulation. 2020 Feb;23(2):177-184. doi: 10.1111/ner.13048. Epub 2019 Sep 16. PMID 31524325
- [Background] Vesper J, Slotty P, Schu S, Poeggel-Kraemer K, Littges H, Van Looy P, Agnesi F, Venkatesan L, Van Havenbergh T. Burst SCS Microdosing Is as Efficacious as Standard Burst SCS in Treating Chronic Back and Leg Pain: Results From a Randomized Controlled Trial. Neuromodulation. 2019 Feb;22(2):190-193. doi: 10.1111/ner.12883. Epub 2018 Nov 19. PMID 30456795
- [Background] Deer TR, Patterson DG, Baksh J, Pope JE, Mehta P, Raza A, Agnesi F, Chakravarthy KV. Novel Intermittent Dosing Burst Paradigm in Spinal Cord Stimulation. Neuromodulation. 2021 Apr;24(3):566-573. doi: 10.1111/ner.13143. Epub 2020 Mar 23. PMID 32202044